CLINICAL TRIAL: NCT00421525
Title: A Phase I/II Study of Immunotherapy With hLL1 Administered Twice Weekly for 4 Consecutive Weeks in Patients With Multiple Myeloma
Brief Title: Phase I/II Study of hLL1 in Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTOCOL: IMMU-115-01
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma; Myeloma, Plasma-Cell; PLASMACYTOMA
Keywords: multiple myeloma; Myeloma, Plasma-Cell; PLASMACYTOMA
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — milatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiple Doses (Other): Multiple Dose levels
  Interventions: Biological: milatuzumab

INTERVENTIONS:
Biological: milatuzumab — twice weekly dosing for 4 weeks, total of 8 doses
  Other Names: CD74; humanized CD74; IMMU-115; hLL1

SUMMARY:
This is a Phase I/II, open-label, multi-center study conducted in patients with recurrent or refractory multiple myeloma who have failed at least two prior standard systemic treatments.

DETAILED DESCRIPTION:
All patients receive hLL1 administered intravenously twice weekly for 4 consecutive weeks. Cohorts of 3-6 patients will receive escalating doses of hLL1 in order to determine the maximum tolerated dose (MTD) for this administration schedule. Up to approximately 30 additional patients will be entered at one or more dose levels at or below the MTD in order to determine the optimal dose for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed, informed consent;
* Male or female, >/=18 years old;
* Meets clinical trial criteria for a diagnosis of multiple myeloma (Appendix 1)
* Stage II or III at study entry by Durie-Salmon staging, with either renal function subclassification (A or B) allowed (Appendix 2).
* Secretory multiple myeloma one or more criteria for measurable disease (serum M protein >1.0 gm/dl measured by serum protein electrophoresis, serum free light chain measurement >200 mg/dl, urinary M protein excretion >200 mg/24 hours);
* Refractory or relapsed to at least two prior standard systemic anti-myeloma treatment regimens;
* Adequate performance status (Karnofsky Scale >/= 60%);
* Life expectancy at least 6 months;
* Adequate hematologic status within 2 weeks before study drug administration:
* Hemoglobin >8.0 g/dL and platelets > 50,000/mm3 (both without transfusion or other hematologic support within 7 days of laboratory testing)
* White blood count (WBC) > 2,000/mm3and absolute neutrophil count (ANC) >1,000/mm3 (both without the use of colony stimulating factors within 7 days of laboratory testing)
* Adequate renal function: serum creatinine < 1.5 x the upper limit of normal (ULN);
* Adequate hepatic function AST or ALT < 2.5 x the ULN; Total bilirubin < 1.5 x the ULN

Exclusion Criteria:

* Pregnant or lactating women.
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study until at least 12 weeks after the last hLL1 infusion;
* Prior chemotherapy, immunotherapy, radiotherapy, plasmapheresis, kyphoplasty, or major surgery within 4 weeks; prior stem cell transplant within 12 weeks; prior treatment with rituximab within 6 months. Must have recovered from all toxicity from prior treatments;
* Prior therapy with other murine, chimeric, human or humanized monoclonal antibodies, unless HAHA tested and negative;
* Prior treatment with any investigational agents within 3 months, unless completed follow-up, off study, and agreed by Sponsor;
* Prior malignancy within 5 years, excluding multiple myeloma, non-melanoma skins cancers and cervical carcinoma in situ;
* Known to be HIV positive, or hepatitis B or C positive;
* Known autoimmune disease or presence of autoimmune phenomena;
* Systemic infection or requiring anti-infectives within 7 days before first dose of study drug;
* Substance abuse or other concurrent medical conditions that, in the investigator's opinion, could confound study interpretation or affect the patient's ability to tolerate or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of hLL1 administered twice weekly for 4 consecutive weeks | first 12 weeks, then over 2 years

SECONDARY OUTCOMES:
The secondary objectives are to obtain information on efficacy, pharmacodynamics, pharmacokinetics, and immunogenicity, and to determine the optimal dose for subsequent studies. | first 12 weeks, then over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (6):
- United States (6):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Center for Cancer Care, Goshen, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Presbyterian Hospital/Cornell Medical Center, New York, New York
  - Hospital University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Sapra P, et al. In vitro and in vivo targeting and therapy of an antibody-drug conjugate (IMMU-110) in B-cell malignancies. (Abstract #3287) Blood 2004; 104/11:898a.
- [Background] Stein R, et al. Therapeutic activity of a new antibody-drug immunoconjugate, IMMU-110, in preclinical studies targeted against multiple myeloma. (Abstract #6535) Proceedings of ASCO 2004; 23:564.
- [Background] Griffiths GL, et al. Promising therapeutic activity of a new drug immunoconjugate, IMMU-110, in a human Burkitt lymphoma model. (Abstract #2381) Blood 2003; 102/11:645a
- [Background] Chang CH, Sapra P, Vanama SS, Hansen HJ, Horak ID, Goldenberg DM. Effective therapy of human lymphoma xenografts with a novel recombinant ribonuclease/anti-CD74 humanized IgG4 antibody immunotoxin. Blood. 2005 Dec 15;106(13):4308-14. doi: 10.1182/blood-2005-03-1033. Epub 2005 Aug 18. PMID 16109781
- [Background] Stein R, Qu Z, Cardillo TM, Chen S, Rosario A, Horak ID, Hansen HJ, Goldenberg DM. Antiproliferative activity of a humanized anti-CD74 monoclonal antibody, hLL1, on B-cell malignancies. Blood. 2004 Dec 1;104(12):3705-11. doi: 10.1182/blood-2004-03-0890. Epub 2004 Aug 5. PMID 15297317
- [Background] Vanama SS, et al. Construction and characterization of a novel ribonuclease immunotoxin consisting of two Ranpirnase (Rap) molecules fused to an internalizing anti-CD74 humanized IgG4 antibody. (Abstract #3289) Blood 2004; 104/11:899a.
- [Background] Burton JD, Ely S, Reddy PK, Stein R, Gold DV, Cardillo TM, Goldenberg DM. CD74 is expressed by multiple myeloma and is a promising target for therapy. Clin Cancer Res. 2004 Oct 1;10(19):6606-11. doi: 10.1158/1078-0432.CCR-04-0182. PMID 15475450
- [Background] Griffiths GL, Mattes MJ, Stein R, Govindan SV, Horak ID, Hansen HJ, Goldenberg DM. Cure of SCID mice bearing human B-lymphoma xenografts by an anti-CD74 antibody-anthracycline drug conjugate. Clin Cancer Res. 2003 Dec 15;9(17):6567-71. PMID 14695162
- [Background] Ong GL, Goldenberg DM, Hansen HJ, Mattes MJ. Cell surface expression and metabolism of major histocompatibility complex class II invariant chain (CD74) by diverse cell lines. Immunology. 1999 Oct;98(2):296-302. doi: 10.1046/j.1365-2567.1999.00868.x. PMID 10540230
- [Derived] Kaufman JL, Niesvizky R, Stadtmauer EA, Chanan-Khan A, Siegel D, Horne H, Wegener WA, Goldenberg DM. Phase I, multicentre, dose-escalation trial of monotherapy with milatuzumab (humanized anti-CD74 monoclonal antibody) in relapsed or refractory multiple myeloma. Br J Haematol. 2013 Nov;163(4):478-86. doi: 10.1111/bjh.12565. Epub 2013 Sep 25. PMID 24112026
- See also: Related Info — http://www.immunomedics.com